CLINICAL TRIAL: NCT01540916
Title: Respiratory Alterations of Acid-base Equilibrium: Acute and Chronic Renal Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 842
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Acute Respiratory Variations of Acid-base Equilibrium
Keywords: acid-base equilibrium; renal system; urinary electrolytes

ARMS (2):
- Hyperventilation (Experimental): Minute ventilation will be increased of about 30% of baseline value, through an increase in respiratory rate
  Interventions: Other: Increase minute ventilation
- Hypoventilation (Experimental): Minute ventilation will be decreased of about 30% of baseline value, through a decrease in respiratory rate
  Interventions: Other: Decrease minute ventilation

INTERVENTIONS:
Other: Increase minute ventilation — Respiratory rate will be increase in order to have a 30% increase of minute ventilation
  Arms: Hyperventilation
Other: Decrease minute ventilation — Respiratory rate will be decrease in order to have a 30% decrease of minute ventilation
  Arms: Hypoventilation

SUMMARY:
Alterations of acid-base equilibrium are very common in critically ill patients. Thus, understanding their pathophysiology and the possible compensatory mechanisms acting in different organs may play an important role in better set the consequent clinical treatment. The lung and the kidney are the two principal actors of such regulations. Although the respiratory response to acid-base alterations is well understood, less information are available for what the renal system is concerned. Such lack of information is partially due to: 1) the historical consideration of the kidney as a "slow" organ, in response to variations in acid-base equilibrium; 2) the lack of a monitoring system to closely assess renal response.

Our group has recently developed a monitoring system aimed at analyzing, in a quasi-continuous and non-invasive manner (every 10 min) the urinary profile in terms of urinary pH and electrolyte concentrations (sodium, potassium, chloride, ammonium).

The investigators hypothesize that the renal system reacts to large as well as to minimal variations of the acid-base equilibrium (especially induced by a variation in the respiratory function) in a very fast way, modifying the urinary concentration (and therefore the urinary excretion) of ammonium and some electrolytes (especially chloride).

DETAILED DESCRIPTION:
Primary aim:

To investigate the acute renal response to respiratory alterations of acid-base equilibrium in order to better understand the underlying physiological mechanisms and to evaluate the validity of a renal monitoring system to indirectly assess the effectiveness of the respiratory function.

Secondary aim:

To collect data on the chronic response of the renal system in patients affected by chronic obstructive pulmonary disease (COPD), as well as on the acute response to acute variation of the chronic respiratory acidosis characterizing patients affected by COPD exacerbation.

Study protol:

Mechanically ventilated patients will undergo controlled variation of the ventilatory setting (hyperventilation vs. hypoventilation) in order to induce a controlled reduction or increase in arterial partial pressure of carbon dioxide (and an increase or reduction of arterial pH), within normal range of pH (7.35 - 7.45) During the variations, urinary concentrations of electrolytes and pH will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of mechanical ventilation
2. Presence of arterial and central venous line
3. Presence of urinary catheter

Exclusion Criteria:

1. acute or chronic renal failure with anuria
2. presence of continuous renal replacement therapy
3. hemodynamic instability
4. less than 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Variations in urinary electrolyte concentrations and pH | From 0 to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Caironi, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Terapia Intensiva Postoperatoria; Rianimazione Generale - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy